CLINICAL TRIAL: NCT02738385
Title: High Intensity Interval- vs Moderate Training on Biomarkers of Endothelial and Cardiovascular Health in Adults: Effect of Postprandial Period
Brief Title: Intensity Training and Cardiovascular Health in Colombian Adults
Acronym: HIIT-Heart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Santo Tomas (Other)
Responsible Party: Principal Investigator, Robinson Ramírez-Vélez, Principal Professor. Center of Studies in Physical Activity Measurements, School of Medicine and Health Sciences, Universidad Santo Tomas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01-1802-2013
Record Dates: First submitted 2016-03-23; First posted 2016-04-14 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Metabolic Diseases
MeSH Terms: conditions — Metabolic Diseases | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Intensity Interval Training (Experimental): Walking on a treadmill 4min at 80-90% peak heart rate and recovery 4 min at 65% peak heart rate until expenditure of 300 kcal until the end of training.
  Interventions: Behavioral: High Intensity Interval Training
- Moderate Intensity Interval Training (Active Comparator): Walking on a treadmill at 60-80% peak heart rate until expenditure of 300 kcal until the end of training.
  Interventions: Behavioral: Moderate Intensity Interval Training

INTERVENTIONS:
Behavioral: High Intensity Interval Training — Exercise will be performed at three sessions per week. All sessions will be supervised by a trained health or exercise professional.
  Arms: High Intensity Interval Training
Behavioral: Moderate Intensity Interval Training — Exercise will be performed at three sessions per week. All sessions will be supervised by a trained health or exercise professional.
  Arms: Moderate Intensity Interval Training

SUMMARY:
Several studies have shown relationship between exercise intensity and improvement cardiometabolic health. It has been suggested that high intensity interval training and also moderate training generate positive effects on metabolic risk factors. For these reasons, it is necessary to clarify which type of training, is more effective to improve cardiometabolic health in latinamerican population.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Interested in improving health and fitness.

Exclusion Criteria:

* Systemic infections.
* Weight loss or gain of >10% of body weight in the past 6 months for any reason.
* Currently taking medication that suppresses or stimulates appetite.
* Uncontrolled hypertension: systolic blood pressure 160 mm Hg or diastolic blood pressure 95 mm Hg on treatment.
* Gastrointestinal disease, including self-reported chronic hepatitis or cirrhosis, any episode of alcoholic hepatitis or alcoholic pancreatitis within past year inflammatory bowel disease requiring treatment in the past year, recent or significant abdominal surgery (e.g., gastrectomy).
* Asthma.
* Diagnosed diabetes (type 1 or 2), fasting impaired glucose tolerance (blood glucose 118 mg/dL), or use of any anti-diabetic medications.
* Currently taking antidepressant, steroid, or thyroid medication, unless dosage is stable (no change for 6 months).
* Any active use of illegal or illicit drugs.
* Current exerciser (>30 min organized exercise per week).
* Indication of unsuitability of current health for exercise protocol (PARQ).
* Any other conditions which, in opinion of the investigators, would adversely affect the conduct of the trial.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in endothelial function as measured by flow-mediated vasodilation (FMD) | Baseline, 2 and 12 weeks immediately after the interventions ends, preceding an 'unhealthy' meal.
  FMD will be measured using the guidelines reported by Corretti et al. The diameter of the brachial artery will be assessed using a high-resolution ultrasound device (Siemens SG-60, USA), equipped with a 7.5 MHz linear array transducer

SECONDARY OUTCOMES:
Change from Baseline in LDL Cholesterol | Baseline, 2 and 12 weeks immediately after the interventions ends, preceding an 'unhealthy' meal.
Change from Baseline in HDL Cholesterol | Baseline, 2 and 12 weeks immediately after the interventions ends, preceding an 'unhealthy' meal.
Change from Baseline in Triglycerides | Baseline, 2 and 12 weeks immediately after the interventions ends, preceding an 'unhealthy' meal.
Change from Baseline in Glucose | Baseline, 2 and 12 weeks immediately after the interventions ends, preceding an 'unhealthy' meal.
Change from Baseline in Heart rate variability | Baseline, 2 and 12 weeks immediately after the interventions ends, preceding an 'unhealthy' meal.
  HRV will be performed according to current recommendations by European Society of Cardiology using an evaluated share-ware
Aortic pulse wave velocity (PWVao) | Baseline, 2 and 12 weeks immediately after the interventions ends, preceding an 'unhealthy' meal.
  PWVao (m s-1) will be performed within 3 to 4 minutes with the oscillometric, occlusive device, the Arteriograph. The measurement will be taken in a supine position and were accepted if the quality indicator of the recordings was within the acceptable range (i.e., if the standard deviation [SD] of the beat-to-beat measured PWVao values was less than 1.1 m/sec).
Change from Baseline in muscular fitness | Baseline, 2 and 12 weeks immediately after the interventions ends, preceding an 'unhealthy' meal.
  Muscular fitness (MF) will be assessed using handgrip test (maximum handgrip strength assessment) using a standard adjustable handle analogue handgrip dynamometer T-18 TKK SMEDLY III®
Change from Baseline in Flexibility using the sit and reach test | Baseline, 2 and 12 weeks immediately after the interventions ends, preceding an 'unhealthy' meal.
  It will be determined using a maximum treadmill exercise test (Precor TRM 885, Italy) following the modified Balke protocol
Change from Baseline in peak uptake of volume of oxygen | Baseline, 2 and 12 weeks immediately after the interventions ends, preceding an 'unhealthy' meal.
Change from Baseline in Blood Pressure | Baseline, 2 and 12 weeks immediately after the interventions ends, preceding an 'unhealthy' meal.
Change from Baseline in Body Mass Index | Baseline, 2 and 12 weeks immediately after the interventions ends, preceding an 'unhealthy' meal.
  BMI will be calculated as the body weight in kilograms divided by the square of the height in meters.
Change from Baseline in Body Mass | Baseline, 2 and 12 weeks immediately after the interventions ends, preceding an 'unhealthy' meal.
Change from Baseline in Quality & satisfaction with life by SF Community - short-form survey (SF-12™) Colombian version | Baseline and 12 weeks immediately after the interventions ends, preceding an 'unhealthy' meal.
Augmentation index (AIx) | Baseline, 2 and 12 weeks immediately after the interventions ends, preceding an 'unhealthy' meal.
  AIx (%) will be performed within 3 to 4 minutes with the oscillometric, occlusive device, the Arteriograph. The measurement will be taken in a supine position and were accepted if the quality indicator of the recordings was within the acceptable range (i.e., if the standard deviation [SD] of the beat-to-beat measured AIx values was less than 1.1 m/sec).

CONTACTS AND LOCATIONS:
Overall Officials: Robinson Ramírez Vélez, Ph.D, Study Director — Universidad del Rosario
Locations (1):
- Robinson Ramírez Vélez Ph.D, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramirez-Velez R, Hernandez-Quinones PA, Tordecilla-Sanders A, Alvarez C, Ramirez-Campillo R, Izquierdo M, Correa-Bautista JE, Garcia-Hermoso A, Garcia RG. Effectiveness of HIIT compared to moderate continuous training in improving vascular parameters in inactive adults. Lipids Health Dis. 2019 Feb 4;18(1):42. doi: 10.1186/s12944-019-0981-z. PMID 30717757
- [Derived] Ramirez-Velez R, Correa-Rodriguez M, Tordecilla-Sanders A, Aya-Aldana V, Izquierdo M, Correa-Bautista JE, Alvarez C, Garcia-Hermoso A. Exercise and postprandial lipemia: effects on vascular health in inactive adults. Lipids Health Dis. 2018 Apr 3;17(1):69. doi: 10.1186/s12944-018-0719-3. PMID 29615070
- [Derived] Ramirez-Velez R, Tordecilla-Sanders A, Tellez-T LA, Camelo-Prieto D, Hernandez-Quinonez PA, Correa-Bautista JE, Garcia-Hermoso A, Ramirez-Campillo R, Izquierdo M. Similar cardiometabolic effects of high- and moderate-intensity training among apparently healthy inactive adults: a randomized clinical trial. J Transl Med. 2017 May 30;15(1):118. doi: 10.1186/s12967-017-1216-6. PMID 28558739
- [Derived] Ramirez-Velez R, Tordecilla-Sanders A, Tellez-T LA, Camelo-Prieto D, Hernandez-Quinonez PA, Correa-Bautista JE, Garcia-Hermoso A, Ramirez-Campillo R, Izquierdo M. Effect of Moderate- Versus High-Intensity Interval Exercise Training on Heart Rate Variability Parameters in Inactive Latin-American Adults: A Randomized Clinical Trial. J Strength Cond Res. 2020 Dec;34(12):3403-3415. doi: 10.1519/JSC.0000000000001833. PMID 28198783